CLINICAL TRIAL: NCT06011083
Title: Calcipotriol /Betamethasone Ointment Versus Fractional CO2 Laser Plus Calcipotriol /Betamethasone Ointment in the Treatment of Plaque Psoriasis: Randomized Comparative Study
Brief Title: Topical Calcipotriol /Betamethasone Ointment in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Hasan Sayed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: psoriasis vulgaris
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Psoriasis Vulgaris; Fractional CO2 Laser
Keywords: psoriasis vulgaris; fractional CO2 laser; Calcipotriol /Betamethasone Ointment
MeSH Terms: interventions — betamethasone-17,21-dipropionate; Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): 20 patients who were treated with Topical Ointment containing Calcipotriol 0.05 mg/gm and Betamethasone dipropionate 0.5 mg/gm twice daily as a monotherapy for 3 months over a selected psoriatic plaque
  Interventions: Drug: Topical Ointment containing Calcipotriol 0.05 mg/gm and Betamethasone dipropionate 0.5 mg/gm
- Group B (Active Comparator): 20 patients who were treated with fractional CO2 laser sessions once per month followed by application of the same Topical Ointment twice daily for 3 months over a similar psoriatic plaque
  Interventions: Drug: Topical Ointment containing Calcipotriol 0.05 mg/gm and Betamethasone dipropionate 0.5 mg/gm; Device: Fractional carbon dioxide (CO2) laser

INTERVENTIONS:
Drug: Topical Ointment containing Calcipotriol 0.05 mg/gm and Betamethasone dipropionate 0.5 mg/gm — using topical ointment containing calcipotriol and betamethasone dipropionate for plaque psoriasis.
Device: Fractional carbon dioxide (CO2) laser — fractional CO2 laser sessions once per month for 3 months over a similar psoriatic plaque
  Arms: Group B

SUMMARY:
comparing the clinical efficacy of topical ointment containing calcipotriol and betamethasone dipropionate used alone with the simultaneous use of fractional carbon dioxide laser and the same topical ointment containing these two ingredients as treatment modalities for plaque psoriasis. Additionally, looking into how both therapy modalities affect individuals with psoriasis in terms of how their quality of life is improved.

DETAILED DESCRIPTION:
Psoriasis is a widespread, persistent papulosquamous skin condition that can affect anyone at any age and places a heavy strain on both the individual and society. It is linked to a number of serious medical disorders, such as cardiometabolic syndrome, depression, and psoriatic arthritis (1).

Patients with psoriasis indicate that the condition interferes with their ability to sleep and rest, limits their everyday activities, particularly their mobility, and stigmatises them and causes problems in their social lives. Additionally, psoriasis can negatively impact mental health. Many psoriasis sufferers struggle with addiction, anxiety, and depression (2, 3).

Topical medicines continue to be the basis of treatment for those with mild psoriasis, and they include topical corticosteroids, vitamin D analogues, calcineurin inhibitors, and keratolytics (4).

For the topical management of mild psoriasis, preparations containing calcipotriol in combination with betamethasone (in the form of betamethasone dipropionate) are available (5). In comparison to the effects of these active substances when given separately, pharmacodynamic investigations demonstrated the synergy between the anti-inflammatory and immunoregulatory actions of calcipotriol and betamethasone dipropionate (6). The synergistic activity of the two drugs is what makes calcipotriol/betamethasone dipropionate combinations successful. Betamethasone impacts inflammatory processes and lessens skin irritation and pruritus following calcipotriol administration, while calcipotriol alters keratinocyte differentiation (7).

Fractional lasers were used in the treatment of dermatological diseases. They create tiny ablation channels in the skin that act as shunts for topically applied medications, particularly those with high molecular weights (8), by ablation of the skin in the form of fractions and splitting laser beams into microbeams (9).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic plaque psoriasis of either sex.
* Aged more than 18 years of age.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with severe skin infection.
* Patients who are under systemic ttt or phototherapy in the last 3 months.
* Immunosuppression or being under any kind of treatment causingabsolute or relative immunosuppression
* History of any bleeding, clotting disorder or using anticoagulants.
* Chronic systemic diseases such as chronic renal failure, hepatic insufficiency, and cardiovascular disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluating the reduction in the severity of the treated psoriatic plaques using Psoriasis severity (TES) score before treatment and after the treatment course in both groups. | 6 month
  Group A included 20 patients who were treated with Topical Ointment containing Calcipotriol 0.05 mg/gm and Betamethasone dipropionate 0.5 mg/gm applied twice daily as a monotherapy for 3 months over a selected psoriatic plaque while Group B included 20 patients who were treated with fractional CO2 laser sessions once per month followed by application of the same topical ointment twice daily for 3 months over a similar psoriatic plaque [as regard anatomical site, size and TES (thickness, erythema, scales) score].
  We used a physician-based, four-point scoring system in which the thickness, erythema, and scale within each plaque was rated from 0 (none) to 3 (severe) to evaluate the changes in the severity of individual psoriatic plaques before treatment and with each visit till the end of the treatment course. The TES score is the sum of the scores given to each individual parameter (thickness, erythema and scale)
to look into how both therapy modalities affect individuals with psoriasis in terms of how their quality of life is improved. | 6 month
  Dermatology Life Quality Index (DLQI) is used for quality of life assessment. The DLQI is a validated, 10-question, self-reported questionnaire. It was done to evaluate the patient's perception of the impact of psoriasis on quality of life before and at the end of the treatment course of both groups (14, 15). The DLQI questionnaire was divided into 6 commonly identified categories. The DLQI was rated on a 4-point scale (0 = not at all to 3 = very much). The highest possible total score for the DLQI is 30 and higher scores indicate more severe impact on quality of life (16). According to the score of the DLQI the impact of psoriasis on QOL is then graded into: no effect at all on patient's life (0-1), small effect (2-5), moderate effect (6-10), very large effect (11-20) and extremely large effect on patient's life (21-30).

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Griffiths CEM, Armstrong AW, Gudjonsson JE, Barker JNWN. Psoriasis. Lancet. 2021 Apr 3;397(10281):1301-1315. doi: 10.1016/S0140-6736(20)32549-6. PMID 33812489